CLINICAL TRIAL: NCT00129610
Title: A Comparative Controlled Study of Virtual Reality Therapy and Cognitive Behavior Therapy in Panic Disorder With Agoraphobia
Brief Title: Study of Virtual Reality Therapy and Cognitive Behavior Therapy in Panic Disorder With Agoraphobia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: 2002.307
Record Dates: First submitted 2005-08-11; First posted 2005-08-12 (Estimated); Last update posted 2007-04-27 (Estimated); Status verified 2007-04

CONDITIONS: Panic Disorder; Agoraphobia
Keywords: Agoraphobia; panic disorder; Virtual Reality Therapy; Cognitive Behavior Therapy; cognition; spatial cognition; PANIC DISORDER WITH AGORAPHOBIA
MeSH Terms: conditions — Panic Disorder; Agoraphobia | interventions — Virtual Reality Exposure Therapy; Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Virtual Reality Therapy
Behavioral: Cognitive Behavior Therapy

SUMMARY:
The study aims at comparing virtual reality therapy (VRT) with a usual cognitive behavior therapy (CBT) program for agoraphobia. A waiting list represents the control condition. The investigators' purpose is to test a pure VRT compared with a pure CBT, as previous works suggest that the combination of the two methods are clinically effective. Patients receive a two-page information leaflet about the trial and sign an informed consent. After the first evaluation, they are randomized, in three centers (Lyon, Paris, Luxemburg), either to VRT (12 sessions) or CBT (12 sessions), or a waiting-list control condition for three months. After three months the waiting list is randomized to VRT or CBT. The follow-up is one year from entry into the active part of the trial.

ELIGIBILITY:
Inclusion Criteria:

* The study includes 90 patients, aged from 18 to 60, with DSM-4 panic disorder with agoraphobia.
* Patients should not be clinically depressed and present a Hamilton Scale of Depression score of less than 18.

Exclusion Criteria:

* Patients with active medication (antidepressants, neuroleptics, mood stabilizers, benzodiazepines, Kava Kava, or hypericum) or street drugs. Minor herbal medicine is tolerated.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90
Dates: Start 2004-01

PRIMARY OUTCOMES:
The response criterion is a decrease of 50% of the agoraphobia subscore on the Fear Questionnaire

SECONDARY OUTCOMES:
Pre-test, post-test, 6 months and one year
Panic Disorder Severity Scale
Agoraphobic cognitions
Panic, phobia, generalized anxiety
Trait State Anxiety Inventory (STAI)
Hamilton Anxiety Scale
Dissociative experiences
Beck Depression Inventory
Quality of Life, handicap
Spatial cognition: Rey's Figure and Rod and Frame test
Therapeutic expectations (pre-test)
Therapeutic relationship (post-test)

CONTACTS AND LOCATIONS:
Overall Officials: Jean COTTRAUX, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Pierre Wertheimer, Bron, France